CLINICAL TRIAL: NCT02287363
Title: Genetic and Morphological Analysis of Thyrotoxic Periodic Paralysis:an Observational Study of Sichuan Individuals in China.
Brief Title: Genetic and Morphological Analysis of Thyrotoxic Periodic Paralysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Haoming Tian, professor, West China Hospital
Other Study IDs: HTian
Record Dates: First submitted 2014-11-05; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Thyrotoxic Periodic Paralysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We intend to draw a 3-5mL whole blood from each participant and extract their genome DNA for genetic analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TPP group: TPP patients(between episodes of paralysis), the inclusion criteria consisted of a certain history of acute limb muscle weakness, hypokalemia and decreased TSH with elevated free FT4, FT3. Subjects who suffered from hyperthyroid myopathy with long term muscle weakness, family periodic paralysis, renal tubular acidosis, hyperaldosteronism, hemiplegia, paraplegia, or any history of other metabolic or traumatic muscular disease were excluded.
  Interventions: Other: No intervention involved
- hyperthyroidism group: Control group, we included subjects with evidence of aberrant thyroid function (decreased TSH, elevated FT4, FT3) without paralysis. Graves' disease(GD) was preferred which required information concerning either increased thyrotrophin receptor antibody(TRAb) level, ophthalmopathy or diffusively enlarged goiter. Individuals with pure thyroid associated ophthalmopathy, history of thyroidectomy due to malignancy or adenoma as well as subacute thyroiditis and pituitary hyperthyroidism were excluded.
  Interventions: Other: No intervention involved

INTERVENTIONS:
Other: No intervention involved — No interventions will be involved since it is an observational study

SUMMARY:
The study aims to analyze the genetic variance between thyrotoxic periodic paralysis (TPP) patients and pure hyperthyroidism individuals. Meanwhile, the investigators also intended to evaluate the morphological difference in effected skeletal muscles and investigate their relation with genetic variance.

DETAILED DESCRIPTION:
Chinese males of their third and forth decades are extremely predisposed to periodic paralysis when they are hyperthyroid. Due to their imbalanced predilection to the disease, genetic variance is considered to be critical to the pathogenesis. In addition, since proximal limb skeletal muscles are the major sites of target, and they are also believed to play a role in the disease generation. Thus, we intend to analyze the genetic and morphological variances between TPP patients and pure hyperthyroidism patients and simultaneously the relation between genetic variance and morphological difference. In this way, we hope to provide evidence for a better understanding of the disease.

ELIGIBILITY:
Inclusion Criteria:

A recent history(within three months) of acute limb muscle weakness, hypokalemia and decreased TSH with elevated free FT4, FT3.

Exclusion Criteria:

Hyperthyroid myopathy with long term muscle weakness, family periodic paralysis, renal tubular acidosis, hyperaldosteronism, hemiplegia, paraplegia, or any history of other metabolic or traumatic muscular disease,

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chinese han population within Sichuan province who is diagnosed with TPP.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Single Nucleotide Polymorphisms | 2 years
skeletal muscle size of biceps brachii and quadriceps femoris | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Haoming Tian, MD., Principal Investigator — West China Hospital